CLINICAL TRIAL: NCT06782607
Title: Clinical Impact of a Multiplex Rapid Diagnostic Pneumonia Panel Testing in Critically-ill Patients with Severe Hospital-acquired Pneumonia, Ventilator-associated Pneumonia and Community-acquired Pneumonia with High Risk of Multidrug Resistant Pathogen
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Adhiratha Boonyasiri, Assistant professor doctor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010/2025
Record Dates: First submitted 2025-01-13; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Infectious Disease of Lung; Molecular Diagnosis; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Pneumonia panel group (Experimental): Pneumonia panel measurement and changing of antimicrobials according to the result of pneumonia panel
  Interventions: Diagnostic Test: Pneumonia Panel by FilmArray
- No Intervention: Standard of care (No Intervention): Standard practice

INTERVENTIONS:
Diagnostic Test: Pneumonia Panel by FilmArray — The Pneumonia Panel comprehensively identifies 33 potential pathogen targets from sputum-like (including endotracheal aspirate) and bronchoalveolar lavage (BAL)-like (including mini-BAL) samples. For 15 of the bacteria, the Pneumonia Panel provides semi-quantitative results, which may help determine whether an organism is a colonizer or a pathogen.
  Arms: Experimental: Pneumonia panel group

SUMMARY:
The objective of the research is to ascertain the influence of a syndromic mutiplex PCR assay (FilmArray) on the management of patients hospitalised in the ICU for severe respiratory disease.

The diagnostic process for pneumonia has become significantly more intricate over the past decade due to the interference of the biological, radiological, and clinical criteria of patients hospitalised in the intensive care unit with the conventional criteria for the diagnosis of severe respiratory diseases. Additionally, patients who are hospitalised in the ICU are at a heightened risk of contracting other associated infections. Consequently, patients are frequently administered antibiotics, whether or not they are effective, as it is challenging to promptly determine the aetiology of their symptoms using conventional methods.

To enhance the diagnostic and therapeutic aspects of their treatment, we implemented a novel syndromic molecular test in our laboratories. This test is designed to expedite and enhance the management of pneumonia and the stewardship of antibiotics. This research will include 80 to 100 adult patients hospitalized in ICU between Feb 2025 and Feb 2027. It will take place within the Siriraj Hospital, Bangkok, Thailand.

DETAILED DESCRIPTION:
Not provided

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received complete information about the research and who have not objected to the use of its data
* Patients with suspected pneumonia infection

Exclusion Criteria: Patients with following conditions;

* Active immediate life-threatening cardiac arrhythmia, defined as ventricular tachycardia and ventricular fibrillation
* Acute cerebral vascular event, including both acute ischemic stroke or intracranial hemorrhage Acute coronary syndrome
* Cardiogenic shock
* Life-threatening gastrointestinal hemorrhage
* Drug overdose
* Advanced-stage cancer with predicted survival less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic decision [Time Frame: 24 hours following the FilmArray results] | 24 hours following the FilmArray results
  Antibiotic prescription modification following the FilmArray results as:
  No prescription No change in antibiotic utilization Antibiotic initiation Antibiotic escalation Antibiotic de-escalation Antibiotic discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stafylaki D, Maraki S, Vaporidi K, Georgopoulos D, Kontoyiannis DP, Kofteridis DP, Chamilos G. Impact of Molecular Syndromic Diagnosis of Severe Pneumonia in the Management of Critically Ill Patients. Microbiol Spectr. 2022 Oct 26;10(5):e0161622. doi: 10.1128/spectrum.01616-22. Epub 2022 Sep 26. PMID 36154180
- [Background] High J, Enne VI, Barber JA, Brealey D, Turner DA, Horne R, Peters M, Dhesi Z, Wagner AP, Pandolfo AM, Stirling S, Russell C, O'Grady J, Swart AM, Gant V, Livermore DM; INHALE Study Group. INHALE: the impact of using FilmArray Pneumonia Panel molecular diagnostics for hospital-acquired and ventilator-associated pneumonia on antimicrobial stewardship and patient outcomes in UK Critical Care-study protocol for a multicentre randomised controlled trial. Trials. 2021 Oct 7;22(1):680. doi: 10.1186/s13063-021-05618-6. PMID 34620213
- [Background] Kosai K, Akamatsu N, Ota K, Mitsumoto-Kaseida F, Sakamoto K, Hasegawa H, Izumikawa K, Mukae H, Yanagihara K. BioFire FilmArray Pneumonia Panel enhances detection of pathogens and antimicrobial resistance in lower respiratory tract specimens. Ann Clin Microbiol Antimicrob. 2022 Jun 4;21(1):24. doi: 10.1186/s12941-022-00512-8. PMID 35659683